CLINICAL TRIAL: NCT02353455
Title: Cells of Monocytic Origin as Surrogate Markers for Individual Drug Effects and Hepatotoxicity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Andreas Benesic, MD (Other)
Collaborators: MetaHeps GmbH (Unknown)
Responsible Party: Sponsor-Investigator, Andreas Benesic, MD, Dr. med., Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Other Study IDs: 055-13
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Drug-induced Disorder of Liver; Adverse Reaction to Drug
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury; Drug-Related Side Effects and Adverse Reactions | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PBMC samples, monocyte derived cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- healthy: donors/patients without liver disease, with and without ongoing drug therapy including buffy coat samples of healthy blood / thrombocyte donors.
  After pseudonymisation a detailed history and clinical data are obtained and blood sampling will be performed . Buffy coats are obtained anonymously.
  Interventions: Procedure: Blood sampling
- prior to therapy: History will be obtained and blood sampling will be performed in patients in whom a drug therapy with a drug with DILI potential is planned.
  Interventions: Procedure: Blood sampling
- iDILI: Patients with clinical suspicion of idiosyncratic drug-induced liver injury. After pseudonymisation a detailed history and clinical data are obtained and blood sampling will be performed.
  Interventions: Procedure: Blood sampling
- non DILI: Patients with other forms of liver injury. After pseudonymisation a detailed history and clinical data are obtained and blood sampling will be performed.
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — In each group a blood sample of approximately 50 mL will be obtained upon study inclusion.

SUMMARY:
Drug metabolism in the liver is subject to large fluctuations (differences between women and men, people of different ethnic backgrounds, children and adults). These large differences are responsible for very different drug effects and side-effects (and especially liver damage caused by drugs) between individuals. Recent scientific findings suggest that blood derived cells can be used to model individual effects of drugs on the liver reflect inter-individual differences. Since liver damage caused by drugs is a diagnosis of exclusion, the aforementioned cells can be used to identify patients that show higher sensitivity to hepatotoxic side-effects and - in case several drugs are involved - identify the causal agent or possible interactions.

DETAILED DESCRIPTION:
Drug-induced liver injury (DILI), especially its idiosyncratic for is often an unpredictable complication of drug therapy. Until now it is very challenging to predict occurrence, severity and outcome of DILI. Previous data provide evidence that cells from peripheral blood may reflect hepatocellular damage (Fannin RD, Hepatology. 2010). Own research could show that peripheral monocytes are capable to obtain several hepatocyte-like functions while maintaining individual characteristics of the donor, especially cytochrome P450 metabolism (Benesic, Gerbes, et al, Lab Invest 2012). This study investigates the effects of potentially hepatotoxic drugs on cells generated from patient blood in comparison to the clinical presentation. Its aim is the evaluation of in vitro tests using monocyte derived cells for diagnosis and exclusion of DILI and the potential to use the patient derived-cells for mechanistic investigations of DILI. 4 groups are investigated: 1) donors without liver disease 2) patients who will start a therapy with DILI-potential; 3) DILI patients; 4) patients with liver injuries other than DILI.

Patient history and clinical data are obtained and a single blood sample will be collected after informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 2 years
* Informed consent given by the patient or in case of inability to give informed consent informed consent of the legally nominated consultee

Exclusion Criteria:

* Anemia requiring blood transfusion
* acute or chronic hepatitis B, C or human immunodeficiency virus infection
* lack of informed consent

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The groups or cohorts will be selected from patients treated at the LMU University Hospital.
  Sampling Method is non-probability sample: patients are invited to volunteer to participate.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-03; Primary Completion 2020-03 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Reflection of individual drug hepatotoxicity in monocyte derived cells | 12 months
  After blood sampling, monocyte derived cells will be generated and tested in vitro for the respective compounds in short term and up to 4 weeks. If possible, the patient will have a clinical follow up during routine care to assess liver injury , course and outcome of the disease when applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander L Gerbes, Prof. MD, Principal Investigator — Liver Center Munich®, Internal Medicine II, Ludwig-Maximilians University Hospital, Campus Grosshadern, Munich; Marchioninistr. 15; D81377 Munich, Germany
Locations (5):
- Gastroenterology, Alfred Health, Melbourne, Victoria, Australia
- Liver Center Munich®, Department of Internal Medicine II, LMU University Hospital, Campus Grosshadern, Munich, Bavaria, Germany
- Chinese University of Hong Kong, Hong Kong, Hong Kong
- Department of Gastroenterology and Hepatology Nagoya University School of Medicine, Nagoya, Japan
- Division of Gastroenterology and Hepatology, Department of Internal Medicine, Korea University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Russo MW, Galanko JA, Shrestha R, Fried MW, Watkins P. Liver transplantation for acute liver failure from drug induced liver injury in the United States. Liver Transpl. 2004 Aug;10(8):1018-23. doi: 10.1002/lt.20204. PMID 15390328
- [Background] Chalasani N, Fontana RJ, Bonkovsky HL, Watkins PB, Davern T, Serrano J, Yang H, Rochon J; Drug Induced Liver Injury Network (DILIN). Causes, clinical features, and outcomes from a prospective study of drug-induced liver injury in the United States. Gastroenterology. 2008 Dec;135(6):1924-34, 1934.e1-4. doi: 10.1053/j.gastro.2008.09.011. Epub 2008 Sep 17. PMID 18955056
- [Background] Watkins PB, Seeff LB. Drug-induced liver injury: summary of a single topic clinical research conference. Hepatology. 2006 Mar;43(3):618-31. doi: 10.1002/hep.21095. PMID 16496329
- [Background] Chalasani N, Bjornsson E. Risk factors for idiosyncratic drug-induced liver injury. Gastroenterology. 2010 Jun;138(7):2246-59. doi: 10.1053/j.gastro.2010.04.001. Epub 2010 Apr 12. PMID 20394749
- [Background] Lee WM. Drug-induced hepatotoxicity. N Engl J Med. 2003 Jul 31;349(5):474-85. doi: 10.1056/NEJMra021844. No abstract available. PMID 12890847
- [Background] Bell LN, Chalasani N. Epidemiology of idiosyncratic drug-induced liver injury. Semin Liver Dis. 2009 Nov;29(4):337-47. doi: 10.1055/s-0029-1240002. Epub 2009 Oct 13. PMID 19826967
- [Background] Zimmerman HJ. Drug-induced liver disease. Drugs. 1978 Jul;16(1):25-45. doi: 10.2165/00003495-197816010-00002. PMID 352664
- [Background] Lee WM, Senior JR. Recognizing drug-induced liver injury: current problems, possible solutions. Toxicol Pathol. 2005;33(1):155-64. doi: 10.1080/01926230590522356. PMID 15805067
- [Background] Fannin RD, Russo M, O'Connell TM, Gerrish K, Winnike JH, Macdonald J, Newton J, Malik S, Sieber SO, Parker J, Shah R, Zhou T, Watkins PB, Paules RS. Acetaminophen dosing of humans results in blood transcriptome and metabolome changes consistent with impaired oxidative phosphorylation. Hepatology. 2010 Jan;51(1):227-36. doi: 10.1002/hep.23330. PMID 19918972
- [Background] Benesic A, Rahm NL, Ernst S, Gerbes AL. Human monocyte-derived cells with individual hepatocyte characteristics: a novel tool for personalized in vitro studies. Lab Invest. 2012 Jun;92(6):926-36. doi: 10.1038/labinvest.2012.64. Epub 2012 Apr 2. PMID 22469698
- [Derived] Weber S, Erhardt F, Allgeier J, Saka D, Donga N, Neumann J, Lange CM, Gerbes AL. Drug-Induced Liver Injury Caused by Metamizole: Identification of a Characteristic Injury Pattern. Liver Int. 2025 Mar;45(3):e70012. doi: 10.1111/liv.70012. PMID 39912769
- [Derived] Weber S, Benesic A, Neumann J, Gerbes AL. Liver Injury Associated with Metamizole Exposure: Features of an Underestimated Adverse Event. Drug Saf. 2021 Jun;44(6):669-680. doi: 10.1007/s40264-021-01049-z. Epub 2021 Feb 27. PMID 33638811
- [Derived] Benesic A, Jalal K, Gerbes AL. Drug-Drug Combinations Can Enhance Toxicity as Shown by Monocyte-Derived Hepatocyte-like Cells From Patients With Idiosyncratic Drug-Induced Liver Injury. Toxicol Sci. 2019 Oct 1;171(2):296-302. doi: 10.1093/toxsci/kfz156. PMID 31407002
- [Derived] Benesic A, Rotter I, Dragoi D, Weber S, Leitl A, Buchholtz ML, Gerbes AL. Development and Validation of a Test to Identify Drugs That Cause Idiosyncratic Drug-Induced Liver Injury. Clin Gastroenterol Hepatol. 2018 Sep;16(9):1488-1494.e5. doi: 10.1016/j.cgh.2018.04.049. Epub 2018 Apr 30. PMID 29723689
- [Derived] Benesic A, Leitl A, Gerbes AL. Monocyte-derived hepatocyte-like cells for causality assessment of idiosyncratic drug-induced liver injury. Gut. 2016 Sep;65(9):1555-63. doi: 10.1136/gutjnl-2015-309528. Epub 2015 Jun 4. PMID 26045135
- See also: Homepage Liver Center Munich — http://www.klinikum.uni-muenchen.de/Lebercentrum/de/index.html